CLINICAL TRIAL: NCT06034366
Title: a Parallel Assignment Prospective, Randomized, Double-blinded, Placebo-controlled Trial to Evaluate the Efficacy of 0.01% Atropine for Near Work-induced Transient Myopia and Myopic Progression
Brief Title: the Efficacy of 0.01% Atropine for Near Work-induced Transient Myopia and Myopic Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: atropine2023
Record Dates: First submitted 2023-08-23; First posted 2023-09-13 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Participants in the study group will use 0.01% atropine (3 ml unit-concentration, preservative-free) once nightly in both eyes for 48 weeks,
  Interventions: Drug: 0.01% atropine
- placebo eye drops (Other): participants in the control group will utilize placebo eye drops (0.9% sodium chloride, 3 ml unit-concentration, preservative-free) once nightly in both eyes for 48 weeks.
  Interventions: Other: 0.9% sodium chloride

INTERVENTIONS:
Drug: 0.01% atropine — 0.01% atropine (3 ml unit-concentration, preservative-free) once nightly in both eyes for 48 weeks,
  Arms: study group
Other: 0.9% sodium chloride — placebo eye drops (0.9% sodium chloride, 3 ml unit-concentration, preservative-free) once nightly in both eyes for 48 weeks
  Arms: placebo eye drops

SUMMARY:
Near work-induced transient myopia (NITM) is an important factor in permanent myopia (PM) development and progression. Atropine eye drop is beneficial in reducing initial NITM and slowing down myopic progression.Participants were randomly assigned in a 1:1 ratio to receive 0.01% atropine or placebo eye drop once nightly bilaterally for one year. Initial NITM, cycloplegic refraction, axial length (AL), best-corrected visual acuity (BCVA), intraocular pressure (IOP), and pupil diameter will be measured at baseline, 4-week, 12-week, 24-week, 36-week, and 48-week. Visual Function Questionnaire was administered at baseline and each follow-up visit. Adverse events also will be monitored and documented at each subsequent follow-up visit. This study investigates the efficacy of 0.01% atropine in the treatment of NITM and its possible association with the progression of refractive change in Chinese myopic children.

DETAILED DESCRIPTION:
Myopia is a common condition that develops primarily during childhood and early adulthood when excessive elongation of the eye results in images of distant objects coming into focus in front of the retina, resulting in blurred distance vision. Myopia is the most common ocular disorder worldwide, with increasing prevalence over the past decades, predominantly in East Asia. Previous studies suggested that environmental factors, such as near-work demands, likely play an important role in myopia development in the younger population.

Near work, a main environmental-based factor in the development and progression of permanent myopia (PM), induced via near work-induced transient myopia (NITM). Compared with PM, NITM refers to the prolonged period required for the accommodation of the eyes to return to a normal level after engaging in a sustained near task. It was proposed some years ago that NITM, which produces minor and chronic retinal defocus, may be one of many possible environmentally-based, myopigenic, contributory factors to permanent myopia.

As a nonselective muscarinic antagonist, atropine eye drops with different concentrations have been reported to slow down the myopic progression in myopes. Recently, a two weeks study assessed the efficacy of a low-concentration of atropine (0.01%) on the initial NITM magnitude among Chinese myopic children. The results suggested 0.01% atropine reduced the initial NITM magnitude. However, the long-term efficacy of 0.01% atropine in treating NITM and the relationship between NITM and refractive change after treatment is still unclear.

This study aimed to investigate the efficacy of 0.01% atropine in treating NITM and its possible association with the progression of refractive change in Chinese myopic children.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 12 years
* Subjects and their guardians agreed to participate in this study
* Best-corrected visual acuity (BCVA) 0.1 (log minimum angle of resolution, LogMAR) or better.
* Initial NITM (spherical equivalent) ≤ -0.25 D
* Cycloplegic refractions ≥ -1.0 D and astigmatism ≤ 2.5 D in both eyes.
* Anisometropia in both eyes ≤ 1.5 D

Exclusion Criteria:

* Children with existing systemic diseases including asthma, collagen disease, immune system disorders, prostate hypertrophy, spastic paralysis, Down's syndrome, severe cardiac, pulmonary, hepatic, and renal dysfunction.
* Patients with glaucoma or high intraocular pressure, ocular inflammatory diseases, strabismus, amblyopia, corneal diseases, diseases of lens, retinal and optic neuropathy
* Regular use of medications that may affect the efficacy of 0.01% atropine, including hairy fruit rutabaga eye drops, tropicamide eye drops, anticholinergic drugs such as pirenzepine and tropicamide, and cholinergic drugs such as carbachol and hairy fruit rutabaga.
* Previous experiences with myopia control therapy.
* A history of allergies to atropine.
* Patients were deemed inappropriate for trial participation by the lead investigator.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Nearwork-induced transient myopia (NITM) in diopter | At baseline, week 4, week 12, week 24, week 36, and week 48
  WAM-5500; Grand Seiko, Japan, will be used to assess the NITM in diopter unit.

SECONDARY OUTCOMES:
Spherical equivalent (SE) in diopter | At baseline, week 4, week 12, week 24, week 36, and week 48
  WAM-5500; Grand Seiko, Japan, will be used to assess the SE of each eye in diopter unit.
Axial length (AL) in millimetre | At baseline, week 4, week 12, week 24, week 36, and week 48
  Zeiss IOL Master 700 will be used to assess the AL of each eye in diopter unit.
25-Item National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) | At baseline, week 4, week 12, week 24, week 36, and week 48
  The NEI-VFQ-25 contains 25 questions: general health, general vision, ocular pain, distance, near tasks, dependency on others, role limitation, mental health, social function, driving, peripheral vision, and color vision difficulty. The answer is converted into a 100-point scale for each question, with 100 being the best and 0 the worst. One or more questions are specific to each subscale; therefore, the subscale score is the average of one or more specific questions. The Chinese version of the NEI-VFQ-25 questionnaire was used

OTHER OUTCOMES:
Safety evaluation of best corrected visual acuity (BCVA) | At baseline, week 4, week 12, week 24, week 36, and week 48
  Best-corrected visual acuity (BCVA) 0.1 (log minimum angle of resolution, LogMAR) chart will be used to assess BCVA of each eye.
Safety evaluation of pupil size | At baseline, week 4, week 12, week 24, week 36, and week 48
  Pupil size in millimetres will be measured using OPD-Scan III, Nidek, Japan.
Safety evaluation of intraocular pressure | At baseline, week 4, week 12, week 24, week 36, and week 48
  Intraocular pressure (IOP) in mmHg using a tonometry.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - He Eye Hospital, Shenyang, Liaoning
  - He Eye Specialist Hospital, Shenyang

IPD SHARING:
Plan to Share IPD: Yes
The study's findings will be shared regardless of the effect's direction. All possible beneficiaries of the research, including patients, carers, family, doctors, advisory boards, and medical boards, will receive trial data. Publications in high-impact, open-access medical journals and talks at national and international medical conferences will serve this purpose.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Baird PN, Saw SM, Lanca C, Guggenheim JA, Smith Iii EL, Zhou X, Matsui KO, Wu PC, Sankaridurg P, Chia A, Rosman M, Lamoureux EL, Man R, He M. Myopia. Nat Rev Dis Primers. 2020 Dec 17;6(1):99. doi: 10.1038/s41572-020-00231-4. PMID 33328468
- [Background] He M, Huang W, Li Y, Zheng Y, Yin Q, Foster PJ. Refractive error and biometry in older Chinese adults: the Liwan eye study. Invest Ophthalmol Vis Sci. 2009 Nov;50(11):5130-6. doi: 10.1167/iovs.09-3455. Epub 2009 Jun 24. PMID 19553618
- [Background] Wong TY, Foster PJ, Hee J, Ng TP, Tielsch JM, Chew SJ, Johnson GJ, Seah SK. Prevalence and risk factors for refractive errors in adult Chinese in Singapore. Invest Ophthalmol Vis Sci. 2000 Aug;41(9):2486-94. PMID 10937558
- [Background] Ciuffreda KJ, Vasudevan B. Nearwork-induced transient myopia (NITM) and permanent myopia--is there a link? Ophthalmic Physiol Opt. 2008 Mar;28(2):103-14. doi: 10.1111/j.1475-1313.2008.00550.x. PMID 18339041
- [Background] Vera-Diaz FA, Strang NC, Winn B. Nearwork induced transient myopia during myopia progression. Curr Eye Res. 2002 Apr;24(4):289-95. doi: 10.1076/ceyr.24.4.289.8418. PMID 12324868
- [Background] Lin Z, Vasudevan B, Ciuffreda KJ, Wang NL, Zhang YC, Rong SS, Qiao LY, Pang CC, Liang YB. Nearwork-induced transient myopia and parental refractive error. Optom Vis Sci. 2013 May;90(5):507-16. doi: 10.1097/OPX.0b013e31828deef1. PMID 23538434
- [Background] Yam JC, Zhang XJ, Zhang Y, Wang YM, Tang SM, Li FF, Kam KW, Ko ST, Yip BHK, Young AL, Tham CC, Chen LJ, Pang CP. Three-Year Clinical Trial of Low-Concentration Atropine for Myopia Progression (LAMP) Study: Continued Versus Washout: Phase 3 Report. Ophthalmology. 2022 Mar;129(3):308-321. doi: 10.1016/j.ophtha.2021.10.002. Epub 2021 Oct 7. PMID 34627809
- [Background] Yam JC, Li FF, Zhang X, Tang SM, Yip BHK, Kam KW, Ko ST, Young AL, Tham CC, Chen LJ, Pang CP. Two-Year Clinical Trial of the Low-Concentration Atropine for Myopia Progression (LAMP) Study: Phase 2 Report. Ophthalmology. 2020 Jul;127(7):910-919. doi: 10.1016/j.ophtha.2019.12.011. Epub 2019 Dec 21. PMID 32019700
- [Background] Guo L, Fan L, Tao J, Hua R, Yang Q, Gu H, Yu S, Li L, Zhao X. Use of Topical 0.01% Atropine for Controlling Near Work-Induced Transient Myopia: A Randomized, Double-Masked, Placebo-Controlled Study. J Ocul Pharmacol Ther. 2020 Mar;36(2):97-101. doi: 10.1089/jop.2019.0062. Epub 2019 Dec 3. PMID 31800355
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Jimenez R, Redondo B, Galan T, Machado P, Molina R, Vera J. Impact of dual-focus soft contact lens wear on near work-induced transient myopia. Clin Exp Optom. 2023 Apr;106(3):296-302. doi: 10.1080/08164622.2022.2029684. Epub 2022 Jan 24. PMID 35073496
- [Background] Chan CW, Wong D, Lam CL, McGhee S, Lai WW. Development of a Chinese version of the National Eye Institute Visual Function Questionnaire (CHI-VFQ-25) as a tool to study patients with eye diseases in Hong Kong. Br J Ophthalmol. 2009 Nov;93(11):1431-6. doi: 10.1136/bjo.2009.158428. Epub 2009 Jun 9. PMID 19515645
- [Background] Miura M, Inomata T, Nojiri S, Sung J, Nagao M, Shimazaki J, Midorikawa-Inomata A, Okumura Y, Fujio K, Akasaki Y, Kuwahara M, Huang T, Nakamura M, Iwagami M, Hirosawa K, Fujimoto K, Murakami A. Clinical efficacy of diquafosol sodium 3% versus hyaluronic acid 0.1% in patients with dry eye disease after cataract surgery: a protocol for a single-centre, randomised controlled trial. BMJ Open. 2022 Jan 31;12(1):e052488. doi: 10.1136/bmjopen-2021-052488. PMID 35105626
- [Derived] Qin G, Chen J, Hu L, Qi Y, Xu L, He W, Yu S, Pazo EE, He X. Protocol for a parallel assignment prospective, randomised, double-blinded, placebo-controlled trial to evaluate the efficacy of 0.01% atropine for near work-induced transient myopia and myopic progression in China. BMJ Open. 2023 Dec 20;13(12):e079833. doi: 10.1136/bmjopen-2023-079833. PMID 38128934